CLINICAL TRIAL: NCT01188863
Title: A Phase 1, Randomized, Open-Label, Three-Way Crossover Study of Two Oral Formulations of LX4211 in Subjects With Type 2 Diabetes Mellitus
Brief Title: Study of Two Oral Formulations of LX4211 in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lexicon Pharmaceuticals (Industry)
Responsible Party: Joel P. Freiman, MD, MPH, Lexicon Pharmaceuticals, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LX4211.1-102-DM; LX4211.102 (Other: Lexicon Pharmaceuticals, Inc.)
Record Dates: First submitted 2010-08-24; First posted 2010-08-26 (Estimated); Last update posted 2011-03-30 (Estimated); Status verified 2011-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol; Fluid Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Solid Oral Dose - 150 mg tablets (Experimental)
  Interventions: Drug: 300 mg LX4211 (150 mg tablets)
- Solid Oral Dose - 50 mg tablets (Experimental)
  Interventions: Drug: 300 mg LX4211 (50 mg tablets)
- Liquid Oral Dose (Experimental)
  Interventions: Drug: 300 mg LX4211 (liquid)

INTERVENTIONS:
Drug: 300 mg LX4211 (150 mg tablets) — Single oral dose of two 150 mg tablets LX4211
  Arms: Solid Oral Dose - 150 mg tablets
Drug: 300 mg LX4211 (50 mg tablets) — Single oral dose of six 50 mg tablets LX4211
  Arms: Solid Oral Dose - 50 mg tablets
Drug: 300 mg LX4211 (liquid) — Single 30 mL dose of liquid oral solution LX4211 (10 mg/mL)
  Arms: Liquid Oral Dose

SUMMARY:
This protocol is intended to compare the effects of both a solid (tablet) and liquid oral dosage form of LX4211 in subjects with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years of age
* Males and females of non-childbearing potential
* Diagnosis of type 2 diabetes mellitus for at least 6 months prior to screening
* Fasting plasma glucose ≤240 mg/dL
* Body mass index <42 kg/sq m
* HbA1c of 7-11%
* C-peptide of ≥1.0 ng/mL
* Ability to provide written informed consent

Exclusion Criteria:

* History of type 1 diabetes mellitus, diabetic ketoacidosis, hyperosmolar nonketonic syndrome, incontinence, or nocturia
* Current use of any blood glucose-lowering agent other than metformin
* Exposure to insulin, thiazide, or loop diuretics within 4 weeks prior to screening
* History of HIV, Hepatitis B, or Hepatitis C
* Surgery within 6 months of screening
* Donation or loss of >400 mL of blood or blood product within 8 weeks prior to start of study
* Use of proteins or antibodies within 12 weeks prior to screening. (Flu shots are allowed.)
* Exposure to any investigational agent or participation in an investigational trial within 30 days of the start of the study
* History of drug or alcohol abuse within 12 months prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2010-09; Primary Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration | Pharmacokinetics samples collected on day of dosing and 24 and 48 hours post-dose (Follow-up).
Time at which maximum observed plasma concentration occurs | Pharmacokinetics samples collected on day of dosing and 24 and 48 hours post-dose (Follow-up).
Half-life of the drug in plasma | Pharmacokinetics samples collected on day of dosing and 24 and 48 hours post-dose (Follow-up).

SECONDARY OUTCOMES:
Plasma glucose | Samples collected on initial visit; Day -15 and Day -5 (Washout); numerous timepoints on Day -1 (Washout) and day of dosing; 24 hours post-dose (Follow-up); and upon discharge.
Urinary glucose excretion | Samples collected on Day -1 (Washout), day of dosing, and 24 and 48 hours post-dose (Follow-up).
Insulin | Samples collected on initial visit; Day -15 and Day -5 (Washout); numerous timepoints on Day -1 (Washout) and day of dosing; 24 hours post-dose (Follow-up); and upon discharge.
Peptide YY | Samples collected on initial visit; Day -15 and Day -5 (Washout); numerous timepoints on Day -1 (Washout) and day of dosing; 24 hours post-dose (Follow-up); and upon discharge.
Glucagon-like Peptide 1 | Samples collected on initial visit; Day -15 and Day -5 (Washout); numerous timepoints on Day -1 (Washout) and day of dosing; 24 hours post-dose (Follow-up); and upon discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Joel P. Freiman, MD, MPH, Study Director — Lexicon Pharmaceuticals, Inc.
Locations (1):
- Lexicon Investigational Site, San Antonio, Texas, United States

REFERENCES:
- [Derived] Zambrowicz B, Freiman J, Brown PM, Frazier KS, Turnage A, Bronner J, Ruff D, Shadoan M, Banks P, Mseeh F, Rawlins DB, Goodwin NC, Mabon R, Harrison BA, Wilson A, Sands A, Powell DR. LX4211, a dual SGLT1/SGLT2 inhibitor, improved glycemic control in patients with type 2 diabetes in a randomized, placebo-controlled trial. Clin Pharmacol Ther. 2012 Aug;92(2):158-69. doi: 10.1038/clpt.2012.58. Epub 2012 Jul 4. PMID 22739142